CLINICAL TRIAL: NCT03017482
Title: Clinical Startup of the 670G Closed Loop Insulin Delivery System
Acronym: 670Gstartup
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Darrell M Wilson, Professor, Stanford University
Other Study IDs: 670Gstartup
Record Dates: First submitted 2017-01-07; First posted 2017-01-11 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Medtronic 670G — This is an open labeled follow up of a clinical startup of a newly approved FDA closed loop insulin delivery system. It is essentially a "prospective" chart review of the clinically startup of a FDA closed loop system and has many elements of a quality improvement project with additional features of:
  * Questionnaires about the utility and impact of the device
  * Use of the device in children younger than the current FDA approval range

SUMMARY:
The purpose of this project is to track initiation and the first year of clinical use of the newly FDA approved 670G closed loop insulin delivery system by patients who have requested this system. Our goal is to evaluate our clinical approach to starting this newly approved system. Since the investigators are only following patients who have already decided to start the 670G, the investigator does not assign specific interventions to the subjects of the study; thus this is a Observational study.

DETAILED DESCRIPTION:
3.1 Initial Procedures After reviewing the patient's interest and eligibility, the investigators will obtain informed consent and assent as appropriate. The investigators will start the clinical process for starting an insulin infusion pump. This typically involves attending a pre-pump class (for those patients naïve to insulin pump therapy) and starting the process to obtain insurance coverage for the 670G system.

The investigators plan to track the insurance approval process, typically the number of calls and faxes required, as well as the result - approved vs not approved.

3.2 Pump Run-in (for those patients new to insulin infusion pumps) For patients who are insulin pump naïve the investigators will start on 670G insulin pump without the glucose sensor activation as per our existing clinical protocol. This may occur at a group visit.

3.3 Initial Visit

During at an initial visit, the following procedures will be performed:

* A clinically obtained HbA1c assessment, typically done via fingerstick and DCA2000 (but any equivalent NGSP-certified point-of-care or laboratory based measurement within 2 weeks prior to enrollment acceptable)
* Collection of medical history information including

  * Demographics (date of birth, gender, race and ethnicity), diabetes history, medical history, concomitant medications
  * Collect data for diabetes devices (eg meters, sensors, pumps)
  * Brief clinical physical exam including vital signs and skin assessment
  * CareLink account creation and sharing of access if this is not already done At this visit, patients will be taught how to insert and use the system glucose sensor.

3.3.1 Initial Week on the 670G System During the following week, the system (with both pump and sensor active) will be active with the PLGS on.

3.4 System Start Visit After the initial PLGS week, patients will be taught, perhaps as a group, the closed loop system and the system activated. (Note: multiple days of system data are required using the pump and sensor prior to the 670G system being capable of delivering additional insulin for hyperglycemia. Therefore, this stage of the start-up is a function of the system requirements.)

3.5 Weekly CareLink Download and Calls For each of the next four weeks, the patient/family will upload data into the CareLink system and the data will be reviewed by a member of the clinical team. Adjustments to system settings will be suggested to the family as clinically appropriate.

3.6 Routine 3, 6, 9 and 12 Month Clinical visits At a routine clinical visits the investigators will obtain an interval medical history, physical examination, collect and review of diabetes management data from all diabetes devices with an eye towards improving glycemic control. The investigators will collect adverse event information regarding severe hypoglycemia and diabetic ketoacidosis. Patients will be advised of suggested changes in pump settings

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not required.
2. Clinically planning to and be able to start the Medtronic 670G closed loop system
3. Age greater than 7.00 years at the initiation of the 670G system
4. Total daily insulin use of great than 8.0 units per day over a 1 week period
5. Willing and able (access to internet from home) to download information into the Medtronic CareLink software

Exclusion Criteria:

* 1) Current or planned pregnancy (for the next 12 months)

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with the clinical diagnosis of type 1 diabetes planning to start the 670G system clinically.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
percent of time patients are on the closed loop system | 6 month
  percent of time patients are on the closed loop system at 6 months after start of closed loop activation with a goal of >70%.

SECONDARY OUTCOMES:
Percent time in range | 6 months
  Percent time in range (70 to 180 mg/dL) "Week 1 before closed loop but with predictive low glucose suspend (PLGS)" vs "Week 24 on full closed loop control."

OTHER OUTCOMES:
Severe Hypoglycemia | 12 months
  Number of severe hypoglycemic events in 12 months on closed loop compared with the up to 12 months before by history before closed loop control
Diabetic Ketoacidosis | 12 months
  Number of diabetic ketoacidosis (DKA) events in 12 months on closed loop compared with the up to 12 months before by history before closed loop control

CONTACTS AND LOCATIONS:
Overall Officials: Darrell M Wilson, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share

REFERENCES:
- [Derived] Lal RA, Basina M, Maahs DM, Hood K, Buckingham B, Wilson DM. One Year Clinical Experience of the First Commercial Hybrid Closed-Loop System. Diabetes Care. 2019 Dec;42(12):2190-2196. doi: 10.2337/dc19-0855. Epub 2019 Sep 23. PMID 31548247